CLINICAL TRIAL: NCT06278246
Title: The Muscarinic Hypothesis of Schizophrenia: an [11C]MK-6884 PET Study Study Protocol
Brief Title: Investigating the Muscarinic System in Schizophrenia Using Positron Emission Tomography
Status: Active, not recruiting | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Other Study IDs: 050/2021
Record Dates: First submitted 2024-02-15; First posted 2024-02-26 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Schizophreniform Disorders
Keywords: Magnetic resonance imaging; Positron emission tomography; Antipsychotic-free
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — arterial blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Schizophrenia: Antipsychotic-free patients with schizophrenia or schizophreniform disorder
  Interventions: Radiation: PET Scan
- Healthy Controls: Healthy controls matched for age, sex, cannabis, and nicotine consumption to the 29 patients
  Interventions: Radiation: PET Scan

INTERVENTIONS:
Radiation: PET Scan — PET scan using the novel [11C]MK-6884 tracer to measure M4R during the antipsychotic-free state

SUMMARY:
Within the schizophrenia population, there are individuals that respond to first-line antipsychotic treatments while others do not. The availability of muscarinic M4 subtype receptors (M4R) may play a role as to whether a person with schizophrenia is responsive to first-line antipsychotics or not. The goal of this observational study is to compare the availability of M4R in antipsychotic-free patients with schizophrenia and matched healthy controls. In addition, M4R availability in schizophrenia patients will be examined in relation to response to first line antipsychotics and clinical and cognitive measures. This study may help better understand antipsychotic resistance in schizophrenia and lead to the development of new treatment options, particularly for cognitive deficits and negative symptoms.

DETAILED DESCRIPTION:
This study is composed of two participant groups. 1) Antipsychotic-free patients with schizophrenia and 2) healthy matched controls. The healthy controls will be matched as closely as possible for age, sex, cannabis, and nicotine consumption to the patient group. All participants will undergo a positron emission tomography (PET) scan to measure the M4R binding with [11C]MK-6884 and examine its relationship with clinical and cognitive measures.

Participants who meet the inclusion and exclusion criteria at screening visit (visit 1) will be enrolled into the study. All participants will undergo a PET scan with the novel tracer [11C]MK-6884 to examine its binding with M4R. The third visit will consist of a MRI scan and cognitive assessments. Participants with schizophrenia will have visit four, which occurs 6 weeks after the first antipsychotic trial, initiated by their treating physician. If the treating physician starts a second antipsychotic trial, then a visit five occurs 6 weeks after the second trial. Both visits four and five involve clinical and cognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

Criteria for both Patients with Schizophrenia and Healthy Controls:

1. Age of 18 years and older
2. Willing to consent to study procedures

Criteria for Patients with Schizophrenia:

1. Inpatients or outpatients ≥18 years of age.
2. DSM-V diagnosis of schizophrenia or schizophreniform disorder confirmed using SCID-5.
3. Capable of consenting to participate in the research study (MacCAT).
4. No exposure to long-acting antipsychotics in the past 6 months and oral antipsychotic-free for at least 2-weeks
5. Deemed suitable to receive first-line antipsychotic treatment as standard of care by the treating physician.

Criteria for Healthy Controls:

1. Absence of history of psychiatric illness using the SCID-5
2. Do not have any first-degree family members with a primary psychotic disorder.
3. Are willing to attend appointments reliably.
4. Are capable of providing consent

Exclusion Criteria:

Participants will be excluded if they meet ANY of the criteria listed below:

1. DSM-V diagnosis of schizoaffective disorder or psychosis not otherwise specified.
2. Unstable medical illness or any concomitant major medical or neurological illness, including a history of seizures and traumatic head injury resulting in a loss of consciousness > 30 minutes that required medical attention.
3. Acute suicidal and/or homicidal ideation.
4. DSM-V substance use disorder (except caffeine and nicotine) within one month prior to study entry.
5. Positive urine drug screen for drugs of abuse at the screening visit (excluding cannabis and/or benzodiazepines).
6. Reporting the chronic use of medication with muscarinic mechanism of action.
7. Pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or any other conditions that would preclude the MRI scan
8. Pregnancy (Note: Females up to age 65 must have negative urine pregnancy test at screening), or breastfeeding.
9. If participation in the study would expose participants to more than the annual radiation dose limit (20 mSv) for human subjects participating in research studies, or if the potential participant already underwent a number of PET scans that, including the PET scans under this protocol, will bring the total to more than 8 PET scans /lifetime. For example, participants known to have already been exposed to radiation through X-rays, CT-scans, or other nuclear medicine procedures during the last year may have already surpassed, or will surpass via study participation, the annual radiation dose limit and thus be excluded.
10. Clinically significant claustrophobia
11. Size of head, neck, and body being unable to fit MRI or PET scanners (e.g. body weight of 350 pounds).
12. Blood or coagulation disorders, or taking anticoagulant medication (not antiplatelet).

Patients with Schizophrenia will also be excluded if they meet ANY of the criteria listed below:

1. Refusal to give consent to investigator to communicate with treating physician for entire duration of the study.
2. Previous clozapine treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Antipsychotic-free patients with schizophrenia or schizophreniform disorder and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
M4 receptor expression | At baseline
  Regional [11C]MK-6884 uptake will be quantified as volume of distribution (VT) and binding potential relative to non-displaceable compartment (BPND), as defined by consensus nomenclature for in vivo imaging of reversibly binding radioligands. Ichise's multilinear analysis (MA1) method will be employed to quantify VT, using arterial blood sampling. The simplified reference tissue model (SRTM) will be used to estimate BPND, using the cerebellum as a reference region.
Clinical Data Statistical Analysis | At baseline and 6 week Follow-up after antipsychotic trial
  Exploratory correlations will be performed between clinical symptoms and whole brain VT within the patient group.

SECONDARY OUTCOMES:
Statistical Analysis of Cognitive Data | At baseline and 6 week Follow-up after antipsychotic trial (only for patient group)
  Correlations will be analyzed between memory performance and dorsal striatal VT within the patient group and healthy control group, respectively. Exploratory correlations will be performed between all other cognitive measures and whole brain VT within each group, separately.
Statistical Analysis of Psychopathological Personality Traits in Health Control Group | At baseline
  Correlations will be performed between trait impulsivity and ventral striatal VT within the healthy control group. Exploratory correlations will be performed between all other personality trait measures and whole brain VT

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Graff, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — https://www.camh.ca/en/science-and-research